CLINICAL TRIAL: NCT03642145
Title: A 52-Week Phase 3B Randomized Open-Label Study Evaluating the Safety and Pharmacokinetics of Emflaza® (Deflazacort) Compared to a Comparable Natural History Control Group in Males Aged ≥2 to <5 Years With Duchenne Muscular Dystrophy (DMD) Followed by a 52-Week Extension Period
Brief Title: A Study of Deflazacort (Emflaza®) in Participants With Duchenne Muscular Dystrophy (DMD)
Acronym: PTCEMF
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Study is no longer necessary given the safety and efficacy of emflaza in this age range has already been established after review of already available data.
Sponsor: PTC Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PTCEMF-GD-003
Record Dates: First submitted 2018-07-10; First posted 2018-08-22 (Actual); Last update posted 2019-06-21 (Actual); Status verified 2019-05

CONDITIONS: Duchenne Muscular Dystrophy
MeSH Terms: conditions — Muscular Dystrophy, Duchenne | interventions — deflazacort

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Arm A: Deflazacort 0.9 mg/kg (Experimental): Participants will receive approximately 0.9 mg/kg deflazacort once daily orally for 52 weeks in Period 1 and for 52 weeks in Period 2. The target dose could be varied +/- 20 percent (%) depending upon the available tablet strengths and change in participant's weight.
  Interventions: Drug: Deflazacort
- Arm B: Deflazacort 0.45 mg/kg (Experimental): Participants will receive approximately 0.45 mg/kg deflazacort once daily orally for 52 weeks in Period 1. Participants will either continue to receive 0.45 mg/kg deflazacort or escalated dose of deflazacort (0.9 mg/kg) once daily orally in Period 2 at the investigator's discretion and in consultation with the caregiver. The target dose could be varied +/- 20% depending upon the available tablet strengths and change in participant's weight.
  Interventions: Drug: Deflazacort
- Natural History Control Group (No Intervention): Control participants matching to the study population as closely as possible, will be used as a comparator to characterize the safety and tolerability of deflazacort.

INTERVENTIONS:
Drug: Deflazacort — Deflazacort tablets will be administered as per schedule and dose specified in respective arms.
  Other Names: Emflaza®
  Arms: Arm A: Deflazacort 0.9 mg/kg; Arm B: Deflazacort 0.45 mg/kg

SUMMARY:
The primary objective of this study is to evaluate the safety of a 0.9 milligrams per kilogram (mg/kg) and 0.45 mg/kg daily dose of deflazacort with a comparable natural history control group after 52 weeks of treatment in males with DMD aged greater than or equal to (>=) 2 to lesser than (<) 5 years.

The study will comprise of 2 periods (Period 1: 52-week safety and pharmacokinetics [PK], and Period 2: 52-week extension). Participants will be randomized in a 1:1 ratio to one of 2 treatment arms: 0.9 mg/kg deflazacort, and 0.45 mg/kg of deflazacort. A historic control group (which should match the study population as closely as possible) will be used as a comparator to characterize the safety and tolerability of deflazacort.

ELIGIBILITY:
Inclusion Criteria:

* In the opinion of the Investigator, the participant and parent(s)/caregiver are capable of complying with protocol requirements.
* The participant's legally acceptable representative signs and dates a written informed consent form and any required privacy authorization prior to the initiation of any study procedures.
* The participant must have a diagnosis of DMD defined by genetic or biopsy confirmation of DMD or have documented, increased serum creatine kinase more than 40 times the upper limit of normal (ULN) and shown phenotypic signs of DMD.
* The participant weighs between 11 kilograms (kg) and 50 kg at screening visit.
* Ability to comply with scheduled visits, oral drug administration, and study procedures.
* The participant is current on childhood vaccinations according to the Center for Disease Control (CDC) recommended immunizations for children from birth through 6 years old. Note: The investigator should discuss timing of receipt of the varicella vaccine with the caregiver prior to initiation of chronic steroid treatment. Administration of live or live attenuated vaccines is not recommended in participants receiving immunosuppressive doses of corticosteroids. Participants whose caregivers decline vaccinations as a matter of personal belief may be included.
* Baseline health is judged to be stable based on medical history, physical examination, laboratory profiles, and vital signs at screening, as deemed by the Investigator.
* The participant is able to ingest the oral tablets either whole or crushed.

Exclusion Criteria:

* The participant has received 4 weeks or more of continuous corticosteroid therapy within 3 months of study screening visit.
* The participant has, in the judgment of the Investigator, clinically significant abnormal clinical laboratory parameters at screening or baseline that may affect safety.
* The participant has, in the judgment of the Investigator, a history or current medical condition that could affect safety including, but not limited to:

  1. Major renal or hepatic impairment
  2. Immunosuppression or other contraindications for corticosteroid treatment
  3. History of chronic systemic fungal or viral infections
  4. Diabetes mellitus or significant glucose intolerance
  5. Idiopathic hypercalciuria
  6. Symptomatic cardiomyopathy Note: Elective surgeries can be discussed with medical monitor.
* The participant has a history of hypersensitivity or allergic reaction to steroids or their formulations including, but not limited to lactose, sucrose, etc.
* The participant has received any drug, including prescription and non-prescription medications, and herbal remedies known to be significant inhibitors and/or inducers of cytochrome P3A4 (CYP3A4) enzymes and/or P glycoprotein (P-gp) 14 days prior to the first dose of study drug.
* The participant has an indication that requires long-term use of strong CYP3A4 inhibitors and/or inducers that would interfere with the pharmacokinetics of deflazacort.
* The participant has received any investigational compound and/or has participated in another clinical study within 30 days prior to study treatment with the exception of observational cohort studies or non-interventional studies.

Ages: 2 Years to 4 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Gender Based: Yes
Enrollment: 0 (Actual)
Dates: Start 2018-10-31 (Actual); Primary Completion 2021-07-31 (Estimated); Study Completion 2021-07-31 (Estimated)

PRIMARY OUTCOMES:
Period 1 and 2: Number of Participants With Treatment Emergent Adverse Events (TEAEs) | 52 weeks
Period 1 and 2: Change From Baseline in Vital Signs and Electrocardiogram (ECG) at Week 52 | Baseline, Week 52
Period 1 and 2: Change From Baseline in the Child Behavior Checklist Score at Week 52 | Baseline, Week 52
Period 1 and 2: Change From Baseline in the Normalized Measure of Bone Density Change (Z-score) for the Dual Energy X-ray Absorptiometry (DEXA) at Week 52 | Baseline, Week 52
Period 1 and 2: Mean Change From Baseline in Height at Week 52 | Baseline, Week 52
Period 1 and 2: Mean Change From Baseline in Body Weight at Week 52 | Baseline, Week 52
Period 1 and 2: Mean Change From Baseline in Height Percentile for Age at Week 52 | Baseline, Week 52
Period 1 and 2: Number of Participants With Clinically Significant Laboratory Tests | 52 weeks

SECONDARY OUTCOMES:
Period 1: Peak Plasma Concentration (Cmax) of Deflazacort | Pre-dose, 0.25, 2, 4, and 6 hours post-dose at Baseline (Week 1) and Week 13
Period 1: Area Under the Curve (AUC) of Deflazacort | Pre-dose, 0.25, 2, 4, and 6 hours post-dose at Baseline (Week 1) and Week 13
Period 1: Volume of Distribution (Vd) of Deflazacort | Pre-dose, 0.25, 2, 4, and 6 hours post-dose at Baseline (Week 1) and Week 13
Period 1: Clearance (CL) of Deflazacort | Pre-dose, 0.25, 2, 4, and 6 hours post-dose at Baseline (Week 1) and Week 13

CONTACTS AND LOCATIONS:
Overall Officials: Francesco Bibbiani, MD, Study Director — PTC Therapeutics